CLINICAL TRIAL: NCT07170254
Title: An Open-Label, Two-Arm, Non-Randomized Clinical Study On The Safety And Efficacy Of Instantaneous CRISPR/Cas9 Gene Editing Therapy For Treating Chinese Patients With HPV-16-Related High-Grade Squamous Intraepithelial Lesions (HSIL)
Brief Title: A Clinical Study on the Evaluation of BD114 for the Treatment HPV-16-Related Cervical HSIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BD-HSIL-114001
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: High-grade Squamous Intraepithelial Lesions (HSIL)
Keywords: High-grade squamous intraepithelial lesions; HPV-16 infection; Gene Editing Therapy
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Gels

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BD114 injection (Experimental): Subgroup 1: Low-dose (n=1)
  * Small lesions (≤5 mm^2): BD114 injection, 0.2 mL
  * Large lesions (>5 mm^2): BD114 injection 0.4 mL
  Subgroup 2: High-dose (n=5)
  * Small lesions (≤5 mm^2): BD114 injection, 0.3 mL
  * Large lesions (>5 mm^2): BD114 injection 0.6 mL
  Interventions: Genetic: BD114VLP, or BD114
- BD114 gel (Experimental): Subgroup 1: Low-dose (n=1)
  * Small lesions (≤5 mm^2): BD114 gel, 0.1 mL
  * Large lesions (>5 mm^2): BD114 gel, 0.2 mL
  Subgroup 2: High-dose (n=5)
  * Small lesions (≤5 mm^2): BD114 gel, 0.2 mL
  * Large lesions (>5 mm^2): BD114 gel, 0.4 mL
  Interventions: Genetic: BD114VLP or BD114 plus Gel

INTERVENTIONS:
Genetic: BD114VLP, or BD114 — CRISPR/Cas9 instantaneous gene editing therapy, called BD114VLP (also BD114) which is a developing product of gene therapy from modified third-generation integrated defective lentivirus, can deliver gRNA/Cas9 ribonucleoprotein complex (RNP). It works to knock out or knock down HPV-16 E6/E7 genes integrated in HSIL cell genome resulting to lesion clearness or regression.
  A single dosing BD114 injection by topical intraepithelial injection of HSIL lesion.
  Arms: BD114 injection
Genetic: BD114VLP or BD114 plus Gel — Genetic: BD114VLP or BD114 plus Gel CRISPR/Cas9 instantaneous gene editing therapy, called BD114VLP (also BD114) which is a developing product of gene therapy from modified third-generation integrated defective lentivirus, can deliver gRNA/Cas9 ribonucleoprotein complex (RNP). It works to knock out or knock down HPV-16 E6/E7 genes integrated in HSIL cell genome resulting to lesion clearness or regression.
  Multiple dosing BD114 gel (BD114 injection :Gel, 1:1) topical application on HSIL, one time every other day, total 5 times (D0, D2, D4, D6, and D8) .
  Arms: BD114 gel

SUMMARY:
This study is intented to evaluate the safety, and tolerability and preliminary efficacy of Instantaneous CRISPR/Cas9 Gene Editing Therapy (BD114 virus-like particle, also BD114) for the treatment of high-grade squamous intraepithelial lesions (HSIL) associated with HPV-16 infection.

DETAILED DESCRIPTION:
This study is an open-label, two-arm, balanced-group, single-dose, non-randomized exploration clinical study. A total of 12 patients with HPV-16 Related HSIL of the Cervix will be enrolled and divided into two arms. Participants in Arm 1 receive topically BD114 intraepithelial injection of lesions, and Participants in Arm 2 receive BD114 gel topical application of lesions, with 6 Participants allocated in each arm. Each study arm is further divided into the low-dose subgroup assigned 1 Participant and the high-dose subgroup assigned 5 Participants. The total study duration for each Participant is 40 weeks (including screening stage). The treatment-emergent adverse events (TEAEs) for safe evaluation, components detection of the BD114 for pharmacokinetics (PK) assessment, histologically lesion regression and virologically HPV-16 clearness for efficacy evaluation are observed and explored during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 25 to 50 years, without childbearing demand;
2. Confirmed histopathological evidence of cervical HSIL (CIN3) at the screening period or within 1 month prior to screening;
3. Confirmed cervical HPV-16 positive by HPV test during the screening period or within 1 month prior to screening, without other high-risk HPV types detected;
4. Complete visibility of both the squamocolumnar junction (SCJ Types 1/2) and the upper margin of acetate-white epithelium or suspected HSIL lesions under colposcopy examine during the screening period or within 1 month prior to screening;
5. No evidence of precancerous lesions or malignancy by endocervical curettage (ECC) ;
6. The biopsy sampling of cervical lesions are performed;
7. Visible residual cervical lesions after screening biopsy;
8. Willing to maintain abstinence or use a highly effective contraceptive method (oral contraceptives, injections, implants, or barrier methods) for women of childbearing potential (WOCBP) from enrollment until Week 36, or her partner undergone surgical sterilization (e.g., vasectomy);
9. Good compliance to protocol-specified procedure in study duration assessed by investigator;
10. Voluntarily participating in the study and willing to provided signed informed consent.

Exclusion Criteria:

1. Positive detection of antibodies or viral test of human immunodeficiency virus (HIV), or hepatitis B virus (HBV), or hepatitis C virus (HCV), or Treponema pallidum (TP) at screening;
2. Confirmed histopathologically epithelial carcinoma, glandular carcinoma or precancerous lesions in the endometrium at screening;
3. Confirmed histopathologically or macroscopically high-grade intraepithelial neoplasia or invasive carcinoma in the vulva, vagina or anus at screening;
4. HSIL with partial location in cervical canal and incomplete colposcopic visualization ;
5. Undergone the treatment for cervical HSIL within 4 weeks prior to screening;
6. Vaccination history of any therapeutic HPV vaccine;
7. Family history of malignancy, or a history/current presence of any malignant tumor;
8. Severe uncontrolled diseases of major organs, including but not limited to: acute myocardial infarction, stroke, liver cirrhosis, severe kidney disease, diabetes mellitus, chronic obstructive pulmonary disease (COPD), hematologic disorders, psychiatric disorders, etc;
9. Pregnant (a positive urine or serum pregnancy test) or lactating women;
10. Participating in another drug or device clinical trial at screening, or participated in one within 3 months prior to screening;
11. The history of any form of gene and/or cell therapy;
12. Drug abuse or alcohol addiction no compliance to protocol-specific procedure;
13. Any other condition unsuitable for participating this study judged by the investigator.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | ~36 weeks
  All AEs and SAEs occurring during the study period (from informed consent signing to Week 36 post-BD114 intervention) were recorded and assessed according to the NCI-CTCAE v5.0 grading system, including their classification by System Organ Class (SOC), severity grade, number of affected Participants, and incidence rates. Gynecological AEs (beyond NCI-CTCAE v5.0 specifications) shall be evaluated by investigators for classification and severity grading according to current clinical guidelines/expert consensus.
Percentage of Participants with No Histologic Evidence of HSIL | Week 24, Week 36
  Cervical tissue biopsies obtained at Week 24 and Week 36 undergo histopathological evaluation, and judge the HSIL Clearance by complete regression or disappear of the original lesions, with clearance rates calculated per the following formula:
  Percentage of Participants with No Histologic Evidence of HSIL (%) = Number of Participants Achieving HSIL Clearance / Total number of Participants treated with BD114 ×100%

SECONDARY OUTCOMES:
Percentage of Participants with No Histologic Evidence of HSIL and No Evidence of HPV-16 | Week 24, Week 36
  Virological HPV-16 assessment was performed using clinically validated type-specific HPV testing kits, meanwhile colposcopy-guided cervical tissue biopsies are histopathologically evaluated. The calculating formula as follow:
  Percentage of Participants with No Histologic Evidence of HSIL and No Evidence of HPV-16 = Number of Participants with No Histologic Evidence of HSIL and No Evidence of HPV-16 / Total number of Participants treated with BD114 ×100%
Percentage of Participants with No Evidence of HPV-16 | Week 24, Week 36
  Histological samples (cervical exfoliated cells) is detected for HPV-16 by real-time fluorescent quantifying PCR technology. The calculating formula as follow:
  Percentage of Participants with No Evidence of HPV-16 = Number of Participants with No Evidence of HPV-16 / Total number of Participants treated with BD114 ×100%
Percentage of Participants with No Evidence of HSIL or LSIL | Week 36
  Cervical biopsies at Week 36 are performed for histopathological evaluation, no histologically evidence of HSIL or LSIL of histological samples are judged as no histology findings of HSIL or LSIL. The calculating formula as follow:
  Percentage of Participants with No Evidence of HSIL or LSIL = Number of Participants with No Evidence of HSIL or LSIL / Total number of Participants treated with BD114 ×100%
Percentage of Participants with No Evidence of HSIL or LSIL and No Evidence of HPV-16 | Week 36
  Cervical biopsies at Week 36 are performed for histopathological evaluation, no histologically evidence of HSIL or LSIL of histological samples are judged as no histology findings of HSIL or LSIL. Histological samples (cervical exfoliated cells) is detected HPV-16 by real-time fluorescent quantifying PCR technology.
  Calculation Formula:
  Percentage of Participants with No Evidence of HSIL or LSIL and No Evidence of HPV-16 = Number of Participants A with No Evidence of HSIL or LSIL and No Evidence of HPV-16 / Total number of Participants treated with BD114 ×100%
Changes in Serum Inflammatory Cytokine (IL-1/IL-6/TNF-α/IFN-γ) Levels Relative to Baseline | Arm 1: at Day 2, Week 1, Week 2, Week 4, Week 12, Week 24, and Week 36. Arm 2: at Day 10, Day 15, Day 22, Day 36, Week 12, Week 24, and Week 36
  Blood samples were collected and analyzed using clinically validated ELISA kits to quantify serum levels of four inflammatory cytokines (IL-1, IL-6, TNF-α, and IFN-γ).
Concentrations of Cas9 Protein and gRNA in Peripheral Blood | Arm 1: at Day 2, Week 1, Week 4, Week 12. Arm 2: at Day 10, Day 15, Day 36, Week 12
  The concentration of Cas9 protein are tested by ELISA and gRNA are detected by qPCR in blood.
Detection of Anti-p24/Cas9 Protein Antibodies in Peripheral Blood | Arm 1: Week 2, Week 4, Week 36. Arm 2: Day 22, Day 36, Week 36
  The detection of anti-p24/Cas9 protein antibodies in blood are performed at scheduled study visits.
Off-Target Analysis | Arm 1: Week 1. Arm 2: Day 15
  Off-Target analysis of cervical biopsy samples is conducted by applying DNA deep sequencing or whole genome sequencing (WGS) to assess BD114-related off-target effects based on the sequencing results.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Hospital of Fudan University, Shanghai, China